CLINICAL TRIAL: NCT05103761
Title: Measuring Low-density Lipoprotein Particle Production and Clearance Rates in Response to Diet-induced Ketosis in Humans
Brief Title: Effect of Diet Induced Ketosis on LDL Turnover Rates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Keto study 21-5376
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-10

CONDITIONS: Ketosis, Metabolic
Keywords: keto diet; ketosis; LDL metabolism; hyperlipidemia; cardiovascular disease
MeSH Terms: conditions — Ketosis; Hyperlipidemias; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the ketogenic diet or the LGIT diet for 8 weeks. Once they complete the first diet, they will go under a washout period for 8 weeks before they start the second diet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketogenic diet (Active Comparator): Diet administered to induce ketosis.
  Interventions: Other: Study diet
- Low glycemic index treatment diet (Placebo Comparator): Diet matched with a ketogenic diet with added carbohydrates to avoid ketosis.
  Interventions: Other: Low glycemic index treatment diet

INTERVENTIONS:
Other: Study diet — A low carbohydrate diet (<20g/day) is administered to achieve diet-induced ketosis.
  Other Names: Nutritional intervention
  Arms: Ketogenic diet
Other: Low glycemic index treatment diet — A diet matched with the study diet with added carbohydrates (40-60g/day) to avoid ketosis.
  Other Names: Control
  Arms: Low glycemic index treatment diet

SUMMARY:
There have been concerning case reports of marked elevations of LDL-c in some individuals consuming a KD and Dr. Lewis has been referred a number of these cases to his lipid clinic, some of whom have had extreme elevations of LDL that mimic familial hypercholesterolemia. These marked elevations of LDLc are unique to a ketogenic diet and far exceed the typical mild elevations seen in those consuming a high fat, low carbohydrate LGIT. The degree of elevation of LDL-c suggests that ketosis per se may impair LDL receptor-mediated LDL particle clearance. This clinical observation is a concerning and clinically important issue since millions of people are consuming this popular diet. There are currently no studies that have examined the mechanism of the LDL-raising effect of a ketogenic diet.

DETAILED DESCRIPTION:
A ketogenic diet (KD) has recently gained popularity amongst the public due to its ability to induce rapid weight loss and for a number of other putative but unproven health benefits. Ketogenic diets also have proven efficacy in resistant cases of seizure disorders. However, due to palatability and adherence issues with KD, alternative diets like the less extreme low glycemic index treatment (LGIT) diet have been effectively used as a seizure disorder treatment option. KD primarily restricts the total amount of carbohydrates in the diet to ≤10% of total caloric intake whereas LGIT primarily restricts high glycemic index foods with total carbohydrates constituting 15% of total energy consumption. While several benefits have been outlined previously, conflicting results have been observed on the effect of diet-induced ketosis on plasma concentrations of the atherogenic low-density lipoprotein cholesterol (LDLc). While some studies showed a significant increase in LDLc with KD treatment, other studies reported the opposite effects with some studies reporting no difference.

Of the studies that reported an increase in LDLc, a review conducted by Chawla et al reported that restricting carbohydrates did not lower LDLc compared to a low-fat diet. In fact, the studies that utilized a low carbohydrate diet reported a significant increase in plasma LDLc concentrations. Similar results were observed by others who reported a significant increase in plasma LDLc within 3 weeks, six months, and 12 months of KD, respectively. Contrary to these findings, Dashti et al reported a significant reduction in plasma LDLc within eight weeks of KD, which remained lower for 24 weeks. Interestingly, in a study conducted by Luukkonen et al, six weeks of KD did not result in any changes in the plasma LDLc. Similar findings were reported by others. With regard to the effect of KD on apoB, limited studies reported that KD increased apoB in the pediatric population but resulted in no change in plasma apoB concentration in adults

. Importantly, there have been concerning case reports of marked elevations of LDL-c in some individuals consuming a KD and Dr. Lewis has been referred a number of these cases to his lipid clinic, some of whom have had extreme elevations of LDL that mimic familial hypercholesterolemia. These marked elevations of LDLc are unique to a ketogenic diet and far exceed the typical mild elevations seen in those consuming a high fat, low carbohydrate LGIT. The investigators speculate that there may be metabolic effects of ketosis per se, independent of the macronutrient composition of the diet that could impair LDL clearance or increase its production. Hence our interest in comparing the effects on LDL metabolism of two low carbohydrate, high-fat diets, differing in their degree of carbohydrate restriction, with and without ketosis. Of course, the investigators cannot completely match the macronutrient composition of the two diets, but the diets will be matched as closely as possible apart from maintaining carbohydrates below or just above the ketogenic threshold, respectively.

Since the popularity of ketogenic diets has increased exponentially amongst the general public in recent years and is commonly used for the treatment of epilepsy, a significant increase in atherogenic LDL-c concentration in those consuming KD could have important public health ramifications. Based on previous literature, at least 1/3rd of the individuals following KD have reported a marked elevation in LDLc levels. Whether this marked elevation in LDLc is due to excess production of LDLc or a defect in clearance is unknown. Due to the complexities and difficulties in quantitating synthesis and clearance rates for LDLc, no studies have been conducted to investigate the changes in LDLc kinetics in response to KD.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 65 years
* Normolipidemic

  * Plasma TG <2.0 mmol/L (~175 mg/dL)
  * HDL >1.0 mmol/L (~40 mg/dL) ) in men or >1.3 mmol/L (50 mg/dL) in women
  * LDLc <4.0 mmol/L (~150 mg/dL)
  * Total cholesterol <5.0 mmol/L (~200 mg/dL)
  * Blood pressure ≤ 140/90 mmHg
  * Fasting plasma glucose ≤ 6.3 mmol/L (125 mg/dL)
  * HbA1c within ≥ 4.0% to ≤ 6.0%
  * Hb > 130
* BMI between 18-30 kg/m2
* Participant agrees to maintain their usual lifestyle and not make any significant changes to activity levels while enrolled in the study
* Cr < 110 umol
* Able to speak and read English
* Agrees to consume each study diet for eight weeks
* Agrees to refrain from alcohol consumption 12 hours before the study

Exclusion Criteria:

* Patients on active treatment using lipid-lowering medications, such as statins, ezetimibe, or bile acid sequestrants
* Use of medications that interfere with protein, carbohydrate, or lipid metabolism (e.g., fish oil capsules)
* Patients who have unstable weight in the past three months (weight loss)
* Patients with a history of gout
* Patients who have had major surgeries
* Abnormal thyroid function or known liver disease
* Patients with chronic kidney disease, decompensated liver disease, unstable cardiac or respiratory disease, or GFR
* Uncontrolled hypertension
* Patients who are pregnant or breastfeeding or peri-menopausal
* Actively attempting to get pregnant or pregnant. Low dose estrogen-containing pill if taken for > 3 months and continued throughout the study is acceptable. Women will be required to use adequate contraception and a pregnancy test will be performed on all women at the time of screening and immediately before each kinetics study.
* Participant has a history of any illness that, in the opinion of the study investigator, might confound the results of the study or pose additional risk to the participant by their participation in the study.
* Abnormal bleeding, frequent headaches, arthritis, stomach problems, SOB, migraines, black outs/fainting, epilepsy, chest pain, asthma
* Participants who consume vegan diet
* Participant consumes excessive amounts of alcohol, defined as >70 g/wk (5 standard drink/wk) for female, and >140 g/wk (10 standard drink/wk) for male.
* One standard drink contains roughly 14 grams of pure alcohol, which is found in: 12 ounces of regular beer, 5 ounces of wine or 1.5 ounces of distilled spirits. Vigorous-intensity physical activity, defined as more than 150 minutes per week of moderate-intensity, or 75 minutes a week of vigorous-intensity aerobic physical activity, or an equivalent combination of both.
* Participant has had major surgery, donated or lost 1 unit of blood (approximately 500 mL) or participated in another investigational study within 4 weeks prior to the prestudy visit.
* Participants have an upcoming special event during the study (wedding, vacation travel, etc.).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
LDL apoB turnover rates | 8 weeks
  The primary objective is to quantitate LDL apoB turnover rates in response to eight weeks of KD-induced ketosis in healthy individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Gary F Lewis, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Tornto General Hospital, UHN, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD with other researchers.